CLINICAL TRIAL: NCT03602404
Title: Estimating the Usual Iodine Intake From Spot Urinary Iodine Concentrations to Obtain the Prevalence of Inadequate or Excess Iodine Intake in School-aged Children and Adults
Brief Title: Estimating Usual Iodine Intake From Spot Urinary Iodine Concentrations
Acronym: ITURN
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Almazov National Medical Research Centre (Other); University of Papua New Guinea (Unknown)
Responsible Party: Principal Investigator, Maria Andersson, Dr., Swiss Federal Institute of Technology
Other Study IDs: ITURN
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Iodine Deficiency
Keywords: Iodine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Spot urine samples Dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- St. Petersburg: School aged children: Generally healthy 9 to 12 years old children
- St. Petersburg: Women of reproductive age: Generally healthy non-pregnant, non-lactating women between 18 and 44 years of age
- Papua New Guinea: School aged children: Generally healthy 9 to 12 years old children

SUMMARY:
The overall objective of this study is to develop a reliable method to obtain habitual iodine intakes from spot urinary iodine concentration (UIC) and to assess the prevalence of inadequate iodine intake in school-age children and women of reproductive age. We will evaluate different methods to estimate iodine intake from UIC and estimate the prevalence of inadequate and excess iodine intake in UIC studies conducted in populations with low, adequate and high iodine intakes using the the established estimated average requirement (EAR)/Tolerable Upper Intake Level (UL) cut-point method.

ELIGIBILITY:
Inclusion Criteria:

* lived in study area >= 12 months
* no reported intake of Amiodarone
* no history of thyroid dysfunction / goiter (past & present)
* no exposure to iodine containing contrast agents within the last 12 months

Second arm: Women aged 18 - 49, exclusion / inclusion criteria apply, plus non-pregnant, non-lactating.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Apparently healthy school-age children and women of reproductive age
Sampling Method: Non-Probability Sample
Enrollment: 1592 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Estimated iodine intake | 17 months
  Estimated daily iodine intake of the study population derived from urinary iodine and creatinine concentrations measured in spot urine samples

SECONDARY OUTCOMES:
Urinary iodine concentration | 17 months
  Measured in spot urine samples and 24 h urine collections
Urinary creatinine concentration | 17 months
  Measured in spot urine samples and 24 h urine collections

CONTACTS AND LOCATIONS:
Locations (2):
- University of Papua New Guinea, Sia, Morobe Province, Papua New Guinea
- Almazov Medical Research Center, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No